CLINICAL TRIAL: NCT02320201
Title: Foot Neuromodulation for Overactive Bladder in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients enrolled for analysis.
Sponsor: Rajeev Chaudhry (Other)
Responsible Party: Sponsor-Investigator, Rajeev Chaudhry, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO14080117
Record Dates: First submitted 2014-12-03; First posted 2014-12-19 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrical stimulation (Experimental): Transcutaneous Electrical Nerve Stimulator (TENS) will be applied to the foot via skin surface electrodes for a minimum of 2 hours per day for 1 week to 20 subjects. Subjects will be required to keep a daily voiding diary for one week before treatment to establish a control, during the treatment week and for one week after treatment. Subjects will also be asked to complete a validated questionnaire prior to treatment, during treatment week and one week after treatment. The primary outcomes of this study are improvement in objective measures of frequency as indicated by voiding diary and subjective symptom improvement based on questionnaire comparison.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulator (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulator (TENS) — Electrical stimulation will be applied to the foot via skin surface electrodes for a minimum of 2 hours per day for 1 week to 20 subjects.

SUMMARY:
To determine the effects of electrical stimulation of the nerves in the foot on overactive bladder conditions in children.

DETAILED DESCRIPTION:
Bladder overactivity in the pediatric population presents a more challenging clinical situation than in adults after failure of medical therapy, as other treatments with proven efficacy such as botulinum injections and interstim sacral nerve stimulators are too invasive for the routine use in children. A non-invasive, effective way to improve overactive bladder in this population would have a great impact on a child's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 5 to 16 years old without any specific neurological disorder or urinary tract infection, clinically diagnosed as idiopathic over active bladder (OAB)
2. Currently having OAB symptoms, i.e. urinary frequency, urgency, or incontinence
3. Having been assessed for and treated if applicable for behavioral etiologies of OAB - holding urine too long, consuming excess caffeine or other bladder irritants.
4. Having been assessed for and treated if applicable for constipation

Exclusion Criteria:

1. Patients with known neurological disorders which may be contributing to OAB symptoms
2. Patients found through history to have significant behavioral causes of OAB including consumption of known bladder irritants and dysfunctional voiding.
3. Patients with chronic constipation who are non-compliant with previous pharmacologic efforts to treat.
4. Patients who are not adequately potty trained
5. Patients who do not tolerate initial stimulation training session in the urology clinic upon enrollment
6. Children with any implantable medical devices such as a pacemaker will be excluded from the study

Note: Any patient currently taking medication such as an anti-muscarinic or a tricyclic antidepressant for overactive bladder at time of enrollment will be eligible to participate and will be continued on their usual medication and dosage throughout the study.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with decreased urinary frequency | 3 weeks
  Foot stimulation decreases urinary frequency measured by a daily voiding diary.

SECONDARY OUTCOMES:
Number of participants with improved over active bladder symptoms | 3 weeks
  Foot stimulation improves OAB symptoms over the course of 3-week period, with foot stimulation applied during the second week measured by a validated symptom survey

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Chaudhry, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh og UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] stimulation in cats. J Urol 2011;186(1):326-30. 2. Chen M, Chermansky C, et al. Electrical stimulation of somatic afferent nerves in the foot increase bladder capacity in healthy human subjects. J Urol. April 2014, 191:1009-1013. 3. Gaziev G, Topazio L, et al. Percutaneous tibial nerve stimulation (PTNS) efficacy in the treatment of lower urinary tract dysfunctions: a systematic review. BMC Urology. 2013, 13:61-72. 4. Sillen U, Arwidsson C, et al. Effects of transcutaneous neuromodulation (TENS) on overactive bladder symptoms in children: A randomized clinical trial. J Pediatr Urol. 2014, in press - accepted 30 March 2014 5. Barroso U, Viterbo W, et al. Posterior tibial nerve stimulation vs parasacral transcutaneous neuromodulation for overactive bladder in children. J Urol. Aug 2013, 190(2):673-677 6. DeGannaro M, Capitanucci ML, et al. Current state of stimulation technique for lower urinary tract dysfunction in children. J Urol. May 2011; 185(5):1571-7. 7. Lordelo P, Teles A, et al. Transcutaneous electrical stimulation in children with overactive bladder: a randomized clinical trial. J Urol. Aug 2010;184(2):683-9. 8. Malm-Buatsi E, NeppleKG, et al. Efficacy of transcutaneous electrical nerve stimulation in children with overactive bladder refractory to pharmacotherapy. Urology 2007. Nov; 70(5):980-3.